CLINICAL TRIAL: NCT01923116
Title: Therapeutic Vaccination Against Human Papillomavirus Type 16 for the Treatment of Anal Intraepithelial Neoplasia in HIV+ Men
Brief Title: Therapeutic HPV-16 Vaccination for the Treatment of Anal Dysplasia
Acronym: VACCAIN-T
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Leiden University Medical Center (Other); ISA Pharmaceuticals B.V. (Industry)
Responsible Party: Principal Investigator, Prof. Jan Prins, Prof. dr. J.M. Prins, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL42802.000.12
Record Dates: First submitted 2013-08-06; First posted 2013-08-15 (Estimated); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Anal Intraepithelial Neoplasia; HIV
Keywords: Anal intraepithelial neoplasia; HIV; HPV; Vaccination; Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HPV-16 vaccine (Experimental)
  Interventions: Drug: HPV-16 vaccine

INTERVENTIONS:
Drug: HPV-16 vaccine — Vaccination with SLP-HPV-01® with or without interferon-a injections.

SUMMARY:
The objective of the study is to assess, in a phase 1/2 study, the safety and efficacy of this synthetic vaccine SLP-HPV-01® in HIV+ men with CD4 counts > 350 x 10E6/l and HPV16-induced intra-anal high-grade AIN (grade 2-3) that failed on, or recurred after previous treatment.

DETAILED DESCRIPTION:
Rationale: Since the introduction of combination antiretroviral therapy (cART), human immunodeficiency virus (HIV)-related morbidity and mortality have considerably decreased. However, as a result of the significantly prolonged life span of HIV-positive patients, new causes of morbidity and mortality have become evident. In particular, anal cancer incidence has increased dramatically in HIV-positive men. Like cervical cancer, anal cancer is causally linked to infections with high-risk papillomaviruses (HPV), and is preceded by cancer precursor lesions: anal intraepithelial neoplasia (AIN). Over 90% of HIV-positive MSM have persisting anal HPV infection, in 88% of patients high-risk HPV is present, and high-grade disease (AIN 2 or 3, HG AIN) is present in 25-52% of all HIV+ MSM. The majority of HG AIN is caused by HPV type 16. As in cervical intraepithelial neoplasia, early diagnosis and treatment of AIN have been advocated to prevent malignancy.

Several treatment options exist for AIN, but success rates are disappointingly low. An alternative strategy might be therapeutic HPV vaccination. In women with vulvar intraepithelial neoplasia (VIN), a condition with a comparable pathogenesis, therapeutic vaccination with a synthetic long-peptide vaccine SLP-HPV-01® , consisting of a mix of long peptides from the HPV-16 viral oncoproteins E6 and E7, was well tolerated, and proved to be effective in a high percentage of women, with a durable response, and induction of HPV-16-specific immunity.

Objective: The objective of the current proposal is to assess, in a phase 1/2 study, the safety and efficacy of this synthetic vaccine SLP-HPV-01® in HIV+ men with CD4 counts > 350 x 10E6/l and intra-anal high-grade, HPV16 positive AIN, who failed on previous treatment.

Study population: HIV-positive MSM with a CD4 count > 350 cells/ul with HPV16-induced intra-anal high-grade AIN (grade 2-3) that was resistant to, or recurred after conventional cauterization or other forms of local treatment.

During the past years the study group in the Academic Medical Center in Amsterdam has built a large cohort of well-characterized HIV-positive patients with histology-proven AIN. Material has been stored of these patients and their lesions. Those patients with AIN resistant to previous treatment will be identified. The causative HPV type will be determined in stored biopsies of these patients, using microdissection (LCM) and in-situ PCR. Only patients with HPV-16-induced lesions (the majority of patients) will be eligible for the current study.

Study design: : The first phase of the study is a dose-response study, with four different dosage schedules (1,5,10; 5,10,20; 10,20,40 and 40,40,40,40 μg of SLP-HPV-01®, administered intradermally with a three-week interval), each dosage schedule with or without the co-administration of pegylated interferon-α (Pegintron 1 μg/kg s.c.) at the day of vaccine administration. Each vaccination schedule is to be tested in 5 patients.

The vaccination schedule that induces in HIV-positive MSM the best HPV16-specific response compared to that of the women with VIN in our previous study, is considered the optimal schedule. The size of this dose group will be increased to a total of 20 patients by treating an additional 15 patients.

Intervention: Patients will be vaccinated 3 or 4 times with a 3-week interval with the SLP-HPV-01® vaccine.

High-resolution anoscopy (HRA) will be performed at inclusion, and repeated at 3, 6,12 and 18 months. The transformation zone will be photographed at each visit. Detailed photos plus biopsies of lesion sites will be obtained. From venous blood samples PBMCs will be obtained before the first (pre), 3 weeks after the first vaccination (post-1), 3 weeks after the second vaccination (post-2), 3 weeks after the third vaccination (post-3) and if applicable 3 weeks after the fourth vaccination (post-4).

Endpoints: The primary clinical end points will be both toxicity/ safety, and the regression of the lesions at 3, 6 and 12 months, as assessed by HRA, with biopsies taken of lesion sites.

Secondary endpoints are regression of lesions at 18 months and HPV16-specific immunity in blood will be measured: i.e. ELISPOT (IFNg) for ex-vivo detection of antigen-specific responses and multiparametric intracellular cytokine/extracellular activation marker staining to determine the type (CD4+ and/or CD8+) and function (activation status and/or cytokines) of T-cells that respond.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age ≥ 18 years
* HIV+ MSM, CD4 count > 350/ul (maximum 3 months before screening visit)
* Biopsy-proven intra-anal high-grade AIN caused by HPV16, resistant to, or recurring after previous treatment with cauterization (or other local treatment), 5FU or imiquimod. A patient is considered resistant to cauterization if after 2 cauterization sessions still lesions are found. A patient is considered resistant to 5FU or imiquimod if after 4 months of weekly (multiple day) application still lesions are found.
* Good performance status (a Karnofsky performance score of ≥60 [on a scale of 0 to 100, with higher scores indicating better performance status])
* Normal pretreatment laboratory blood values as described previously. This means: Leukocytes >3 x 109/L, lymfocytes >1 x 109/L, trombocytes >100 x 109/L and hematocrit >30%.

Exclusion Criteria:

* Immunosuppressive medication or other diseases associated with immunodeficiency
* Life expectancy < 1 year
* History of anal carcinoma
* IFN-α criteria (see SmPC): severe cardiac, thyroid, hepatic or central nervous system disease, including severe depression in the past.
* Previous HPV vaccination
* Currently treated with IFN-α against hepatitis C

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-08; Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Safety/ toxicity of the HPV-16 vaccine in HIV+ MSM | up to 18 months
  Monitoring for spontaneous adverse events and injection-site reactions will be done weekly for three weeks after each vaccination. Clinical assessments and laboratory tests (routine hematology and chemistry) will be performed before the second and third vaccination and thereafter every 3 months for a total of 18 months of follow-up. Adverse events are graded according to version 3.0 of the Common Terminology Criteria for Adverse Events (CTCAE), which grades events on a scale of 1 to 5, with higher grades indicating greater severity.

SECONDARY OUTCOMES:
Regression of intra-anal high grade AIN lesion | Primary outcome: 3, 6, 12 months. Secondary: 18 months.
  High resolution anoscopy is performed to monitor the AIN lesions. Biopsies will be obtained of suspected lesions. Complete response is defined as histological resolution of AIN, partial response is defined as regression from high grade to low grade AIN. In case of persisting high grade AIN, a partial response is defined as a decrease in lesion size of 50% or more.

OTHER OUTCOMES:
HPV16-specific immunity in blood | 3 weeks after the 1st, 2nd and 3rd vaccination
  In order to assess the systemic changes in immunity, which are induced by vaccination we will examine venous blood samples by using peripheral blood lymphocytes that are tested by a set of complementary T-cell assays: i.e. proliferation (LST), cytokine production (IFNg, TNFa, IL-4, IL-5, IL-10, and IL-2) as well as by ELISPOT (IFNg) for ex-vivo detection of antigen-specific responses and by multiparametric intracellular cytokine/extracellular activation marker staining to determine the type (CD4+ and/or CD8+) and function of T-cells that respond.
  A vaccine-induced response is defined as a 3-fold increase compared to the pre-vaccination result.
Regression of peri-anal high grade AIN lesions | 3, 6, 12 and 18 months
  High resolution anoscopy is performed to monitor the AIN lesions. Biopsies will be obtained of suspected lesions. Complete response is defined as histological resolution of AIN, partial response is defined as regression from high grade to low grade AIN. In case of persisting high grade AIN, a partial response is defined as a decrease in lesion size of 50% or more.

CONTACTS AND LOCATIONS:
Overall Officials: Jan M Prins, prof, MD, infectiologist, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Henry JC de Vries, prof, MD, dermatologist, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Amsterdam, North Holland, Netherlands